CLINICAL TRIAL: NCT02145962
Title: Application of Extremely Low Frequency Electromagnetic Fields in the Cicatrization of Ulcers With Diabetic Origin as a Method of Preventive and Complementary Treatment
Brief Title: Open Multi-center Safety & Efficacy Study of Low Frequency Magnetic Fields to Treat Unresponsive Diabetic Foot Ulcers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Autonomous University of Morelos (Other)
Collaborators: Universidad Autonoma de Nuevo Leon (Other); Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Luis Enrique Alberto Cañedo Dorantes, Research Professor, MD PhD, Autonomous University of Morelos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELF-MF-2006-001; AVANCE-C2005-219 (Other: National Council for Science and Technology Mexico (CONACYT))
Record Dates: First submitted 2014-05-16; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Neuropathic Diabetic Ulcer - Foot
Keywords: diabetic foot ulcer healing; magnetic therapy; safety and efficacy; wound care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Forearm tissue exposure with ELF-MF (Active Comparator): This study arm should include subjects with diabetic foot ulcers recruited at the medical services site of the Autonomous University of Nuevo Leon, Monterrey, Mexico. These study patients should receive treatment in the forearm region.
  Interventions: Device: Forearm tissue exposure with ELF-MF
- Thorax tissue exposure with ELF-MF (Active Comparator): This study arm should include subjects with diabetic foot ulcers recruited at the IMSS Regional General Hospital N. 1 and Servicios de Salud de Morelos, Cuernavaca, Mexico. These study patients received treatment in the thorax region.
  Interventions: Device: Thorax tissue exposure with ELF-MF

INTERVENTIONS:
Device: Forearm tissue exposure with ELF-MF — The treatment was delivered 2 hours/day, 2 times/week and consisted of sinusoidal oscillating magnetic fields of 120 Hz using a solenoid, with nominal field amplitude of approximately 0.6-0.8 mT (6-8 Gauss) RMS at the center of the stimulation system. The amount of blood exposed to the therapeutic ELF-MF using the forearm device is approximately 30 ml/min or 3.6 lt/session.
  Arms: Forearm tissue exposure with ELF-MF
Device: Thorax tissue exposure with ELF-MF — The treatment was delivered 25 minutes/day, 2 times/week and consisted of 120 Hz using a quasi-Helmholtz coil configuration, with nominal field amplitude of approximately 0.6-0.8 mT (6-8 Gauss) RMS at the center of the stimulation system. The amount of blood exposed to the therapeutic ELF-MF using the thorax device should be approximately 6,500 ml/min or 162.5 lt/session, which is approximately 45 times more blood volume stimulation per unit of time compared with the Forearm exposure system.
  Arms: Thorax tissue exposure with ELF-MF

SUMMARY:
An open multicenter trial to document the efficacy and safety of two therapeutic Extremely Low Frequency Magnetic Fields stimulation devices to promote wound healing of Diabetic Foot Ulcers.

DETAILED DESCRIPTION:
An open multi center trial to document the systemic effects and safety of Extremely Low Frequency Electromagnetic Fields (ELF-MF) stimulation on healing of Diabetic Foot Ulcers (DFU). The study will be performed in two sites: Monterrey, Nuevo Leon, with patients from Medical Services of the Autonomous University of Nuevo León, and Cuernavaca, Morelos with patients from Regional General Hospital of Cuernavaca N. 1 IMSS, and Health Services of Morelos.

Two ELF-MF investigational exposure systems will be used to stimulate blood at different anatomical regions to enhance wound healing upon peripheral blood mononuclear cell migration to the ulcer site. a) In Monterrey, Nuevo Leon, where DFU subjects should be exposed at either forearm with a sinusoidal oscillating magnetic field of 120 Hz with nominal ELF-MF amplitude of approximately 0.6mT-0.8mT (6-8 Gauss) RMS 2 hours/day, 2 times/week. and b) In Cuernavaca, Morelos, where DFU subjects would be exposed at the thorax with a stimulation system in a quasi-Helmholtz configuration, for 25 minutes/day, 2 times/week to a sinusoidal oscillating magnetic field of 120 Hz, with nominal ELF-MF amplitude of approximately 0.6mT-0.8mT (6-8 Gauss) RMS. Treatment period for both groups will be 14.2 weeks or upon a complete healing. In each treatment session, evolution of ulcer healing should be recorded photographically.

Efficacy and adverse effects will be searched for during treatment, short-term (<1 year), and long-term follow-up in both groups (up to 7 years).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 20 years old
* Presence of diabetic foot ulcers resistant to medical and/or surgical treatment
* Medical care prior to admission.

Exclusion Criteria:

* Pregnant women
* Cancer diagnosis
* BMI > 3
* Non-diabetic leg ulcers
* Infected wounds
* Skin autoimmune disease
* Vasculitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Diabetic foot ulcer healing time | 14.2 weeks or upon complete ulcer healing
  Healing time was defined as the period (in days) required for the completion of ulcer closure when applying electromagnetic field treatment. Treatment period end-point was 14.2 weeks or upon complete healing according to clinical inspection.

SECONDARY OUTCOMES:
Adverse events | Two periods: 1 year and up to 7 years
  After treatment, follow-ups were performed to assess short-term (<1 year) and long-term safety (up to 7 years) after treatment. Adverse events were also assessed and defined as: a) Ulcer recurrences in the same site, b) Damage to an organ, c) Development of cancer or any other disease states possibly associated to the use of Extremely Low Frequency Magnetic Fields treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Canedo Dorantes, MD, PhD, Principal Investigator — Autonomous University of Morelos; Guillermo Cabrera Alvarez, MD, Study Chair — Instituto Mexicano del Seguro Social; Rogelio Salinas Dominguez, MD, Study Chair — Universidad Autonoma de Nuevo Leon
Locations (2):
- Mexico (2):
  - Hospital General Regional No. 1 "Ignacio García Tellez" IMSS, Cuernavaca, Morelos
  - Medical Services of the Autonomous University of Nuevo Leon, Monterrey, Nuevo León

REFERENCES:
- [Background] Canedo-Dorantes L, Garcia-Cantu R, Barrera R, Mendez-Ramirez I, Navarro VH, Serrano G. Healing of chronic arterial and venous leg ulcers through systemic effects of electromagnetic fields [corrected]. Arch Med Res. 2002 May-Jun;33(3):281-9. doi: 10.1016/s0188-4409(02)00357-0. PMID 12031635